CLINICAL TRIAL: NCT05060952
Title: Synovial Fluid Calprotectin Lateral Flow Test for the Diagnosis of Prosthetic Joint Infection
Brief Title: Calprotectin in Chronic Prosthetic Joint Infection
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Technical University of Munich (Other)
Responsible Party: Principal Investigator, Christian Suren, Associate Professor, Technical University of Munich
Other Study IDs: 26/19 S-SR
Record Dates: First submitted 2021-09-19; First posted 2021-09-29 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Prosthetic Joint Infection; Prosthetic Infection; Arthroplasty Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- PJI: Patients with septic arthroplasty failure
  Interventions: Diagnostic Test: Calprotectin Lateral Flow Test
- Aseptic: Patients with aseptic causes of arthroplasty failure
  Interventions: Diagnostic Test: Calprotectin Lateral Flow Test

INTERVENTIONS:
Diagnostic Test: Calprotectin Lateral Flow Test — Semiquantitative point of care photometric assay for the calprotectin level in joint fluid aspirate

SUMMARY:
A bacterial infection of an artificial joint is a serious complication that often requires additional surgery to exchange the arthroplasty. It is also difficult to recognize an infected joint, as the symptoms caused by the infection are very similar to those of other problems with arthroplasties, such as loosening of the implant. To improve the ability to diagnose prosthetic joint infections, this study compares the levels of calprotectin, a specific inflammatory protein, in the joint fluid of infected joints and joints with other complications. The underlying hypothesis is that the level of calprotectin in infected joints is significantly higher, thus facilitating the diagnosis of prosthetic joint infection.

ELIGIBILITY:
Inclusion Criteria:

* scheduled arthroplasty exchange for any of the following reasons:
* infection
* loosening
* instability
* malalignment
* periprosthetic fracture

Exclusion Criteria:

* acute prosthetic joint infection

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with painful or failed arthroplasty of the hip or knee joint scheduled for partial or complete arthroplasty exchange.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of synovial fluid calprotectin | Intraoperatively
  The level of synovial fluid calprotectin measured in joint fluid aspirate as a diagnostic test for prosthetic joint infection. The accuracy is calculated by comparing its results with the International Consensus Meeting (ICM) on prosthetic joint infection criteria of 2018.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Orthopedics and Sports Orthopedics, Klinikum rechts der Isar, Technical University Munich, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No